CLINICAL TRIAL: NCT00646048
Title: A Phase I Evaluation of the Safety of the TriVascular Stent-Graft System in the Treatment of Abdominal Aortic Aneurysms
Acronym: AAA IDE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Colleen Holthe, Boston Scientific
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2106
Record Dates: First submitted 2008-03-26; First posted 2008-03-28 (Estimated); Results first posted 2011-01-19 (Estimated); Last update posted 2011-01-28 (Estimated); Status verified 2011-01

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Abdominal Aortic Aneurysm; AAA; TriVascular Stent-Graft System; Stent-Graft
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): This arm is for patient that receive the TriVascular Stent-Graft System.
  Interventions: Device: TriVascular Stent-Graft System

INTERVENTIONS:
Device: TriVascular Stent-Graft System — TriVascular Stent-Graft System

SUMMARY:
This study was a prospective observational study examined the safety of the TriVascular AAA Stent-Graft System in the elective treatment of patients with abdominal aortic aneurysms. Specifically, the study will evaluate the safety of the TriVascualr AAA Stent-Graft System, evaluate the ability to deliver the Tri-Vascular AAA Stent-Graft System to the desired location within the aorta, and evaluate the ability of the TriVascular AAA Stent-Graft to exclude the abdominal aortic aneurysm.

ELIGIBILITY:
Inclusion Criteria:

* Male or infertile female
* Have signed an informed consent form.
* Are considered an appropriate candidate for open surgical repair of an abdominal aortic aneurysm.
* at least one of the following: Abdominal aortic aneurysm >= 4.5 cm in diameter; aneurysm has increased in size by 0.5cm in last 6 months; maximum diameter of aneurysm exceeds 1.5 times the transverse dimension of an adjacent normal aortic segment; saccular aneurysm larger than 3 cm.
* Have patent iliac or femoral arteries that allow endovascular access to the aneurysmal site with a 17F Delivery Catheter.

Exclusion Criteria:

* A dissecting, acutely ruptured, or leaking aneurysm, or an acute vascular injury due to trauma.
* A need for emergent surgery.
* contraindication to undergoing angiography.
* A Thoracic aortic aneurysm that requires treatment.
* Presence of thrombus or atheroma in proximal aortic neck covering > 50% of the endoluminal surface.
* Presence of diffuse atherosclerotic disease in either common iliac artery that reduces the iliac artery diameter to <7mm.
* Congenital abnormalities in which the placement of the stent-graft will cause occlusion of major arterial flow. Such abnormalities should be evaluated(e.g. angiography or CT) prior to treatment.
* Unstable angina
* Morbid obesity or other clinical conditions that severely inhibit x-ray visualization of the aorta.
* Connective tissue disease (e.g., Marfan's or Ehlers-Danlos syndrome.)
* Hypercoagulable state.
* Contraindication for anticoagulation.
* Acute renal failure.
* Active systemic infection.
* less than 18 years of age.
* Life expectancy less than 1 year.
* Current, or anticipated participation within 1 year, in another research study involving an investigational device or new drug (with the exception of participation in the Lifeline Registry of Endovascular Therapy).
* Other medical, social, or psychological issues that in the opinion of the investigator preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-02; Primary Completion 2004-11 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Grady, PhD, Study Director — Boston Scientific Corporation
Locations (7):
- United States (7):
  - Harbor UCLA Medical Center, Torrance, California
  - Georgetown University Pasquerilla Healthcare, Washington D.C., District of Columbia
  - University of Florida - Shands Hospital, Gainesville, Florida
  - Miami Cardiac & Vascular Institute Baptist Hospital, Miami, Florida
  - Albany Medical College, Albany, New York
  - University of Pennsylvania Medical Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Shadyside Hospital, Pittsburgh, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- TriVascular Stent Graft: This arm is for patients that receive the TriVascular Stent-Graft System. The TriVascular Stent Graft Systems was designed to treat patients with Abdominal Aortic Aneurysms(AAA). The stent-graft was designed to provide an alternate intraluminal blood conduit and isolate the aneurysm from the blood flow.
Period: Overall Study
Arm/Group | TriVascular Stent Graft
Started | 43
Completed | 27
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | TriVascular Stent Graft
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 73.1 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 36
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Without a Device Related Adverse Events Within 1 Month of the Study Procedure.
Description: Device related adverse events included, but were not limited to: Stent Graft Migration, Vessel dissection or perforation, stent graft occlusion, branch vessel occlusion, aneurysm rupture.
Time Frame: 1 month
Measure: Number; unit: Participants
Arm/Group | TriVascular Stent Graft
Number analyzed (Participants) | 43
Participants | 36

2. Primary Outcome: Number of Participants Without a Type I, III, and/or IV Endoleak at 1 Month Follow-up Identified by Computed Tomography (CT).
Description: A Type I endoleak is a persistent perigraft channel of blood flow that develops due to inadequate or ineffective seal at the graft ends (attachment zones). A Type III endoleak occurs in the midgraft region due to leakage through a defect in the graft fabric or between the segments of a multisegmental graft. A Type IV endoleak is seen on completion of angiography or subsequent contrast studies as any blush of contrast that is presumed to emanate from blood diffusion across the porous graft fabric or through small holes in the graft cause by sutures or stent struts.
Time Frame: 1 month
Measure: Number; unit: Participants
Arm/Group | TriVascular Stent Graft
Number analyzed (Participants) | 43
Participants | 0

3. Secondary Outcome: Number of Participants Who Achieve Technical Success of the Stent Graft System.
Description: Technical success was defined as successful introduction of the delivery catheter into the arterial system at the time of the study procedure and successful delivery/deployment of the stent graft system to the intended location with the absence of device related surgical conversion and intra-operative mortality. Device related surgical conversion is defined as the inability to deliver or deploy the stent graft system, then subsequently surgically treating the patient.
Time Frame: Post procedure
Measure: Number; unit: Participants
Arm/Group | TriVascular Stent Graft
Number analyzed (Participants) | 43
Participants | 42

ADVERSE EVENTS:
Time Frame: Baseline through 5 year follow-up.
Arm/Group | TriVascular Stent Graft
Serious Adverse Events (participants affected / at risk) | 35/43
Other Adverse Events (participants affected / at risk) | 33/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TriVascular Stent Graft (N=43)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Angina pectoris (Cardiac disorders) | 3 (3)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Cardiac disorder (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 4 (7)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ventricular hypokinesia (Cardiac disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Catheter site related reaction (General disorders) | 2 (2)
Death (General disorders) | 1 (1)
Ulcer (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Bacteriuria (Infections and infestations) | 1 (1)
Catheter site cellulitis (Infections and infestations) | 1 (1)
Catheter site infection (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (2)
Endocarditis bacteraemia (Infections and infestations) | 1 (1)
Enterococcal bacteraemia (Infections and infestations) | 1 (1)
Gangrene (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Stent related infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Arterial injury (Injury, poisoning and procedural complications) | 3 (3)
Device breakage (Injury, poisoning and procedural complications) | 7 (7)
Device failure (Injury, poisoning and procedural complications) | 6 (7)
Device migration (Injury, poisoning and procedural complications) | 2 (2)
Device occlusion (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1)
Medical device complication (Injury, poisoning and procedural complications) | 1 (2)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Stent occlusion (Injury, poisoning and procedural complications) | 8 (8)
Stent-graft endoleak (Injury, poisoning and procedural complications) | 8 (11)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Thrombosis in device (Injury, poisoning and procedural complications) | 3 (3)
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Laboratory test abnormal (Investigations) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Refractory anaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 3 (3)
Transient ischaemic attack (Nervous system disorders) | 2 (3)
Mental status changes (Psychiatric disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal artery stenosis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic surgery (Surgical and medical procedures) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1)
Aorto-duodenal fistula (Vascular disorders) | 1 (1)
Arterial thrombosis limb (Vascular disorders) | 1 (1)
Embolism (Vascular disorders) | 1 (1)
Haemorrahage (Vascular disorders) | 2 (3)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 5 (5)
Iliac artery occlusion (Vascular disorders) | 1 (1)
Iliac artery thrombosis (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 2 (2)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1)
Vascular pseudoaneurysm (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TriVascular Stent Graft (N=43)
Catheter site haematoma (General disorders) | 3 (3)
Catheter site related reaction (General disorders) | 3 (3)
Device breakage (Injury, poisoning and procedural complications) | 12 (12)
Stent-graft endoleak (Injury, poisoning and procedural complications) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Intermittent claudication (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other